CLINICAL TRIAL: NCT00746941
Title: A Randomized, Rater-Blinded Study to Explore the Effect of Mefloquine in Subjects With Progressive Multifocal Leukoencephalopathy (PML)
Brief Title: Study to Explore the Effect of Mefloquine in Participants With Progressive Multifocal Leukoencephalopathy (PML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Primary endpoint not achieved
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111JC101
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: PML; Human Polyomavirus JC; HIV; Central Nervous System Disease; Mefloquine; JC Virus
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal; Central Nervous System Diseases | interventions — Mefloquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local standard of care (No Intervention): All participants received local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  Participants in this treatment arm had the option of adding 250 mg mefloquine by mouth at Week 4 (Day 28) or Week 8 (Day 56) daily for 3 days, and then weekly through Week 24.
- Local standard of care plus mefloquine 250 mg (Experimental): All participants received local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  Participants received 250 mg mefloquine by mouth on Days 0, 1, and 2 and then weekly through Week 24.
  Interventions: Drug: mefloquine

INTERVENTIONS:
Drug: mefloquine — 250 mg orally each day for 3 days and then weekly up to 6 months.
  Other Names: Lariam®; Mephaquin®; Mefliam®
  Arms: Local standard of care plus mefloquine 250 mg

SUMMARY:
The primary objective of the study was to explore whether mefloquine can delay or stop progression of progressive multifocal leukoencephalopathy (PML) as measured by JC virus (human polyomavirus or JCV) deoxyribonucleic acid (DNA) levels in cerebrospinal fluid (CSF). The secondary objective of the study was to explore whether mefloquine can delay or stop progression of PML based on neurological deterioration, magnetic resonance imaging (MRI) measures of brain lesion evolution or the formation of new lesions, and mortality.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PML confirmed by detection of JCV DNA in CSF.
* Onset of PML symptoms within 6 months prior to study.

Key Exclusion Criteria:

* Other opportunistic infection of the central nervous system.
* Current severe illness or any other conditions that, in the opinion of the Investigator, would make the subject unsuitable for enrollment.
* Active severe mental illness (e.g., depression, anxiety, psychosis, and schizophrenia).
* Hypersensitivity to mefloquine, quinine, or quinidine, or to any component of these drugs.
* Current treatment with quinine, quinidine, chloroquine, or halofantrine.

Note: Other protocol-defined criteria may also apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
- Research Site, São Paulo, Brazil
- Germany (3):
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Berlin
  - Research Site, Hamburg
- Research Site, Milan, Italy
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

REFERENCES:
- [Result] Clifford DB, Nath A, Cinque P, Brew BJ, Zivadinov R, Gorelik L, Zhao Z, Duda P. A study of mefloquine treatment for progressive multifocal leukoencephalopathy: results and exploration of predictors of PML outcomes. J Neurovirol. 2013 Aug;19(4):351-8. doi: 10.1007/s13365-013-0173-y. Epub 2013 Jun 4. PMID 23733308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve sites enrolled participants prior to study termination.
Pre-assignment Details: Participants were initially randomized in a 1:1 ratio to the local standard of care arm (represented below as 3 treatment arms depending on Week 4 and Week 8 decisions) or the local standard of care plus mefloquine 250 mg arm.
Groups:
- Local Standard of Care: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  These participants received only local standard of care throughout the study; they did not choose to add 250 mg mefloquine at Week 4 (Day 28) or Week 8 (Day 56).
- Local Standard of Care; Mefloquine at Week 4: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  These participants chose to add 250 mg mefloquine by mouth at Week 4 for 3 days and then weekly through Week 24 to their local standard of care treatment.
- Local Standard of Care; Mefloquine at Week 8: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  These participants chose to add 250 mg mefloquine by mouth at Week 8 for 3 days and then weekly through Week 24 to their local standard of care treatment.
- Local Standard of Care Plus Mefloquine 250 mg: Participants were randomized to receive local standard of care (which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital) and 250 mg mefloquine by mouth on Days 0, 1, and 2 and then weekly through Week 24.
Period: Overall Study
Arm/Group | Local Standard of Care | Local Standard of Care; Mefloquine at Week 4 | Local Standard of Care; Mefloquine at Week 8 | Local Standard of Care Plus Mefloquine 250 mg
Started | 7 | 5 | 5 | 20
Completed | 0 | 1 | 3 | 7
Not Completed | 7 | 4 | 2 | 13
Not completed — Death | 2 | 0 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 2
Not completed — Other, reason not provided | 2 | 4 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Standard of Care | Local Standard of Care; Mefloquine at Week 4 | Local Standard of Care; Mefloquine at Week 8 | Local Standard of Care Plus Mefloquine 250 mg | Total
Number analyzed (Participants) | 7 | 5 | 5 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (20.56) | 41.6 (11.37) | 47.4 (10.06) | 48.1 (9.4) | 47.2 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5 | 10
  Male | 6 | 3 | 3 | 15 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 4 | 9
  White | 6 | 3 | 3 | 16 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Disease history [Number; unit: participants] — Participants were stratified into the following groups
  * HAART-naïve stratum: human immunodeficiency virus (HIV) -positive participants who developed PML in the absence of highly active anti-retroviral therapy (HAART) were placed in this stratum.
  * History of HAART stratum: HIV-positive participants who developed PML while on HAART were placed in this stratum.
  * HIV-negative stratum: All participants who were HIV-negative were placed in this stratum.
  participants
    HIV positive: HAART Naive | 3 | 5 | 3 | 13 | 24
    HIV positive: History of HAART | 1 | 0 | 1 | 3 | 5
    HIV negative | 3 | 0 | 1 | 4 | 8
JVC Titer at Screening [Number; unit: participants] — JC virus (human polyomavirus) titer prior to study randomization.
  participants
    <= 50 copies/mL | 0 | 0 | 0 | 4 | 4
    > 50 copies/mL | 7 | 5 | 5 | 15 | 32
    Missing | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in JC Virus (JCV) Load in Cerebrospinal Fluid (CSF)
Description: Change from baseline to Week 4 in JC viral load in CSF is expressed as log10 copies/mL. Negative values indicate a reduction in viral load.
  Only participants with measurable baseline values are included. Post-baseline values of 'Below the Limit of Quantification' or 'Below Limit of Detection' or 'Negative' were set to 50. Log10 (50) = 1.699
Time Frame: Day 0 (baseline), Week 4
Population: Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
  Participants with undetectable CSF JCV load at baseline were not included in the efficacy analysis. All other enrolled participants were included in the efficacy analysis if values for Week 4 were available.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Local Standard of Care: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 13 | 14
log10 copies/mL | -0.2424 (0.83556) | -0.0675 (1.52685)
Statistical Analysis 1: Comparison: Local Standard of Care vs Local Standard of Care Plus Mefloquine 250 mg; Test type: Superiority or Other; p = 0.7132, Student's t-test

2. Primary Outcome: Change From Baseline to Week 8 in JC Virus (JCV) Load in Cerebrospinal Fluid (CSF)
Description: Change from baseline to Week 8 in JC viral load in CSF is expressed as log10 copies/mL. Negative values indicate a reduction in viral load.
  Only participants with measurable baseline values are included. Post-baseline values of 'Below the Limit of Quantification' or 'Below Limit of Detection' or 'Negative' were set to 50. Log10 (50) = 1.699
Time Frame: Day 0 (baseline), Week 8
Population: Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
  Participants with undetectable CSF JCV load at baseline were not included in the efficacy analysis. All other enrolled participants were included in the efficacy analysis if values for Week 8 were available.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 4 | 10
log10 copies/mL | -0.2843 (0.68666) | -0.3455 (0.93960)
Statistical Analysis 1: Comparison: Local Standard of Care vs Local Standard of Care Plus Mefloquine 250 mg; Test type: Superiority or Other; p = 0.9086, Student's t-test

3. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in the Expanded Disability Status Scale (EDSS) Score
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death) was calculated. Negative change scores indicate improvement.
Time Frame: Day 0 (baseline), Week 4 and 8
Population: Participants with values at the time frames being measured. EDSS was not required for participants who had physical or cognitive impairments that limited their ability to perform the assessment.
  Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
units on a scale
  Week 4 (n=12, 21) | 0.79 (1.054) | 0.50 (1.129)
  Week 8 (n=7, 16) | 0.71 (1.868) | 0.88 (1.360)

4. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in Karnofsky Performance Status (KPS) Index Score
Description: The KPS Index classifies participants' functional impairment. KPS can be used to compare effectiveness of different therapies and to assess the prognosis in individual participants. KPS was recorded on an 11-point scale (0, 10, 20, 30, 40, 50, 60, 70, 80, 90, and 100.) where '0=Dead' and '100=Normal, no complaints, no evidence of disease'. The lower the KPS score, the worse the survival for most serious illnesses. The KPS index is subdivided into 3 categories: incapacitated (0 to 40), self-care (50 to 70), and normal activity (80 to 100).
  Negative change from baseline scores indicate improved prognosis.
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: Participants with values at the time frames being measured. Participants with undetectable CSF JCV load at baseline by the central laboratory were not included in the efficacy analysis.
  Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
units on a scale
  Week 4 (n=12, 21) | 0.00 (14.771) | -8.10 (12.891)
  Week 8 (n=7, 16) | -10.0 (26.46) | -10.6 (19.14)

5. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in Symbol Digit Modalities Test (SDMT)
Description: The SDMT is a simple substitution task. The test gives participants 90 seconds to pair specific numbers with given geometric figures as a measure for screening cognitive impairment. The total score is the total number of correctly completed boxes in the time allowed. The test score range is from 0 (worst outcome) to 110 (best outcome).
  Negative change from baseline scores indicates a worsening outcome.
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: Participants with values at the time frames being measured. SDMT was not required for participants who had physical or cognitive impairments that limited their ability to perform the assessment.
  Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
units on a scale
  Week 4 (n=6,8) | 4.00 (6.723) | -1.50 (3.780)
  Week 8 (n=3,6) | 1.7 (10.12) | 3.8 (6.43)

6. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in Participants' Neurological Function Using a Visual Analog Scale (VAS)
Description: Participants rate their neurological function on a scale of 100 mm line, where the 0 end of the scale indicates poor neurological function and 100 indicates excellent neurological function. VAS was not required for participants who had physical or cognitive impairments that limited their ability to perform the assessment.
  Negative change from baseline scores indicates a worsening outcome.
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: Participants with values at the time frames being measured. VAS was not required for participants who had physical or cognitive impairments that limited their ability to perform the assessment.
  Local standard of care participants who added mefloquine at Week 4 or Week 8 were counted as being dosed under both treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
units on a scale
  Week 4 (n=9,16) | 8.9 (29.14) | -0.7 (33.71)
  Week 8 (n=4,13) | 26.3 (49.00) | 3.5 (23.87)

7. Secondary Outcome: Participants With Gadolinium (Gd)-Enhanced Lesions at Baseline, Week 4 and Week 8 as Seen on Magnetic Resonance Imaging (MRI) Scans of Participants' Brains
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
participants
  Week 0 (n=15,21) | 8 | 8
  Week 4 (n=12,12) | 5 | 8
  Week 8 (n=5,11) | 1 | 7

8. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in T1 Lesion Volume as Seen on Magnetic Resonance Imaging (MRI) Scans of Participants' Brains
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 mm^3
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
log10 mm^3
  Week 4 (n=12,11) | 0.1407 (0.20345) | 0.1631 (0.22523)
  Week 8 (n=5,11) | 0.0248 (0.12425) | 0.1029 (0.26502)

9. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in T2 Lesion Volume as Seen on Magnetic Resonance Imaging (MRI) Scans of Participants' Brains
Time Frame: Day 0 (baseline), Week 4, Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 mm^3
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
log10 mm^3
  Week 4 (n=12,11) | 0.1704 (0.22012) | 0.1619 (0.17501)
  Week 8 (n=5,10) | 0.1738 (0.21454) | 0.1050 (0.23429)

10. Secondary Outcome: Participants Who Died Within 6 Months
Description: The death event is counted under the treatment arm relative to adding mefloquine to the treatment regimen.
Time Frame: Day 1 up to 6 months
Population: Safety population: All participants who enrolled in the study and were dosed, and who have at least 1 post-baseline safety assessment.
  The death event is counted under the treatment arm relative to adding mefloquine to the treatment regimen.
Measure: Number; unit: participants
Groups:
- Local Standard of Care Plus Mefloquine 250 mg: Participants were randomized to receive local standard of care (which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital) and 250 mg mefloquine by mouth on Days 0, 1, and 2 and then weekly through Week 24.
  Also includes participants who were randomized to receive local standard of care (only) and added mefloquine at Week 4 or Week 8.
Arm/Group | Local Standard of Care | Local Standard of Care Plus Mefloquine 250 mg
Number analyzed (Participants) | 17 | 30
participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Day 1 to Month 6
Description: Because participants were primarily patients with HIV/Acquired Immunodeficiency Syndrome (AIDS), SAEs considered to be AIDS-Defining Events (ADEs) were exempt from SAE reporting and were collected on a specific case report form instead of being captured as SAEs. However, any ADE that resulted in death did not qualify for an SAE exemption.
Groups:
- Local Standard of Care: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  Participants who chose to add mefloquine at Weeks 4 or 8 to their standard of care treatment are counted in this treatment arm until the time of switching to mefloquine treatment.
- Local Standard of Care; Mefloquine at Week 4: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  Participants who chose to add mefloquine at Week 4 to their standard of care treatment are counted in this treatment arm once mefloquine treatment started.
- Local Standard of Care; Mefloquine at Week 8: Participants were randomized to receive local standard of care, which may have included any treatment or procedure that the Investigator would normally use in the treatment of a PML patient at their study site or hospital.
  Participants who chose to add mefloquine at Week 8 to their standard of care treatment are counted in this treatment arm once mefloquine treatment started.
Arm/Group | Local Standard of Care | Local Standard of Care; Mefloquine at Week 4 | Local Standard of Care; Mefloquine at Week 8 | Local Standard of Care Plus Mefloquine 250 mg
Serious Adverse Events (participants affected / at risk) | 5/17 | 1/5 | 3/5 | 13/20
Other Adverse Events (participants affected / at risk) | 12/17 | 4/5 | 5/5 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Local Standard of Care (N=17) | Local Standard of Care; Mefloquine at Week 4 (N=5) | Local Standard of Care; Mefloquine at Week 8 (N=5) | Local Standard of Care Plus Mefloquine 250 mg (N=20)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 2 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 3
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Local Standard of Care (N=17) | Local Standard of Care; Mefloquine at Week 4 (N=5) | Local Standard of Care; Mefloquine at Week 8 (N=5) | Local Standard of Care Plus Mefloquine 250 mg (N=20)
Headache (Nervous system disorders) | 0 | 2 | 1 | 4
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 2
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 2
Apallic syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 2 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 1
Extensor plantar response (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 1
Disarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0 | 3
Anogenital warts (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 1 | 0 | 0
Pyomyositis (Infections and infestations) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal mucosal hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 1 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1 | 1
Mucosal membrane hyperplasia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Infusion site haematoma (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 2
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysphemia (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1
Scotoma (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Inflammation of lacrimal passage (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Skin turgor decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 2 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0
Neurological examination abnormal (Investigations) | 1 | 0 | 0 | 0
Prealbumin decreased (Investigations) | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Phlebolith (Vascular disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hilar lymphaedenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1
Dilatation ventricular (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dennie-Morgan fold (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Immune reconstitution syndrome (Immune system disorders) | 2 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
From ongoing analysis, it became clear, based on conditional power calculations, that the study would not reach its primary endpoint, a decrease of JC viral load in CSF with mefloquine treatment; therefore, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 45 to 60 days as agreed within their clinical trial agreement to review any manuscript for a proposed publication and must delay publication for up to an additional 60 to 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.